CLINICAL TRIAL: NCT06170723
Title: A Phase 1, 2-Part, Open-Label, Fixed-Sequence Study to Evaluate the Effects of Itraconazole, Food, and pH, on the Single Dose Pharmacokinetics of BMS-986368 in Healthy Participants
Brief Title: A Study to Assess the Effects of Itraconazole, Food, and pH on the Drug Levels of BMS-986368 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM045-1002
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Healthy Participants
Keywords: BMS-986368; Itraconazole; Famotidine; Food Effect; Healthy Volunteers
MeSH Terms: interventions — Itraconazole; Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: BMS-986368 - Fasted (Experimental)
  Interventions: Drug: BMS-986368
- Part 1: Itraconazole - Fasted (Experimental)
  Interventions: Drug: Itraconazole
- Part 1: BMS-986368 with Itraconazole - Fasted (Experimental)
  Interventions: Drug: BMS-986368; Drug: Itraconazole
- Part 2: BMS-986368 - Fasted (Experimental)
  Interventions: Drug: BMS-986368
- Part 2: BMS-986368 - Fed (Experimental)
  Interventions: Drug: BMS-986368
- Part 2: Famotidine, followed by BMS-986368 - Fasted (Experimental)
  Interventions: Drug: BMS-986368; Drug: Famotidine

INTERVENTIONS:
Drug: BMS-986368 — Specified dose on specified days
  Arms: Part 1: BMS-986368 - Fasted; Part 1: BMS-986368 with Itraconazole - Fasted; Part 2: BMS-986368 - Fasted; Part 2: BMS-986368 - Fed; Part 2: Famotidine, followed by BMS-986368 - Fasted
Drug: Itraconazole — Specified dose on specified days
  Arms: Part 1: BMS-986368 with Itraconazole - Fasted; Part 1: Itraconazole - Fasted
Drug: Famotidine — Specified dose on specified days
  Arms: Part 2: Famotidine, followed by BMS-986368 - Fasted

SUMMARY:
This 2-part study will evaluate the effect of coadministration of a Cytochrome P450, family 3, subfamily A (CYP3A) inhibitor, itraconazole (Part 1), and a high-fat/high-calorie meal and a modified gastric pH (Part 2), on the single dose drug levels of BMS-986368 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 18.0 kilograms per meter squared (kg/m^2) to 33.0 kg/m^2, inclusive.

Exclusion Criteria:

* Personal or first-degree family history of clinically significant psychiatric disorder, including, but not limited to, schizophrenia, psychosis, bipolar disorder, generalized anxiety disorder, obsessive-compulsive disorder, and post-traumatic stress disorder. Situational depression, or anxiety in the past, may be enrolled at the discretion of the investigator.
* Participant has an active or prior history of stroke, chronic seizures, or major neurological disorders or has first-degree family relative who was diagnosed with these disorders below the age of 65 years.
* Participant has a history of syncope and/or symptomatic orthostatic hypotension in the year prior to Day 1.

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 11 days
Area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration (AUC[0-T]) | Up to 11 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC[INF]) | Up to 11 days

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 41 days
Number of participants with physical examination abnormalities | Up to 17 days
Number of participants with vital sign abnormalities | Up to 17 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 17 days
Number of participants with clinical laboratory abnormalities | Up to 17 days
Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to 17 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html